CLINICAL TRIAL: NCT00050973
Title: Randomized Phase III Trial Comparing Targretin Capsules/Cisplatin/Vinorelbine Versus Cisplatin/Vinorelbine in Chemotherapy-Naive Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Evaluation of Efficacy, Safety and Tolerability of Targretin Capsules in Patients With Advanced or Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L1069-49; NCT00030927 (obsolete NCT alias)
Record Dates: First submitted 2002-12-31; First posted 2003-01-03 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2008-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Targretin; Retinoid; Bexarotene
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bexarotene

INTERVENTIONS:
Drug: bexarotene

SUMMARY:
This study evaluates the use of Targretin capsules (bexarotene) in combination with standard chemotherapy for the treatment of metastatic Non-Small Cell Lung Cancer (NSCLC) in patients who have not yet received chemotherapy for their lung cancer.

DETAILED DESCRIPTION:
This study evaluates the use of Targretin capsules (bexarotene) in combination with Cisplatin and Vinorelbine for the treatment of metastatic non-small cell lung cancer in patients who have not yet received chemotherapy for their lung cancer. Every patient receives a platinum-containing chemotherapy every four weeks for at least four chemotherapy cycles (approximately four months). Half of the patients are randomly assigned to receive Targretin capsules once daily in addition to the chemotherapy. The other half is randomized to receive a standard platinum-containing chemotherapy without Targretin capsules.

ELIGIBILITY:
Patients must have:

* Pathologic (histologic or cytologic) confirmation of NSCLC
* Stage IIIB with malignant pleural effusion or Stage IV disease
* At least one measurable or evaluable NSCLC lesion that has not been previously irradiated unless radiation therapy was more than three weeks prior to entry in the study and the lesion has been shown to have progressed subsequent to the radiation therapy
* ECOG performance status 0 or 1
* Adequate organ system function
* Fasting serum triglycerides that are within the age-adjusted normal range (or normalized with appropriate intervention such as antilipid therapy prior to the initiation of Targretin capsule therapy).

Patients must be able to complete at least four cycles of combination chemotherapy (i.e., approximately four months)

Patients must not have had:

* Brain metastasis
* Prior chemotherapy for NSCLC
* Prior platinum-based chemotherapy for any indication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Primary Completion 2004-11 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mack Mabry, M.D., Study Director — Ligand Pharmaceuticals
Locations (77):
- United States (20):
  - Brookwood Medical Center, Birmingham, Alabama
  - Southern Arizona VA Healthcare System, Tucson, Arizona
  - Arroyo Research Inc., Pasadena, California
  - Desert Hematology-Oncology Medical Group, Inc., Rancho Mirage, California
  - University of Florida, Gainsville, Florida
  - New Hope Cancer Center, Hudson, Florida
  - Veterans Affairs Medical Center, Miami, Florida
  - Bay Area Cancer Consultants, Palm Harbor, Florida
  - Northwest Medical Specialists, Arlington Heights, Illinois
  - Jayne Gurtler, M.D., APMC, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - St. Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - SUNY Downstate Medical Center, Brooklyn, New York
  - VA Western New York Health Care System, Buffalo, New York
  - Hematology-Oncology Associates, Toledo, Ohio
  - Tariq Mahmood, Midwest City, Oklahoma
  - University Oncology & Hematology Associates, Chattanooga, Tennessee
  - Marshfield Medical Research Foundation, Marshfield, Wisconsin
  - Medical Associates Health Centers, Menomonee Falls, Wisconsin
- Australia (8):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Southern Medical Daycare Centre, Wollongong, New South Wales
  - Burnside War Memorial Hospital, Toorak Gardens, South Australia
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Border Medical Oncology, Wodonga, Victoria
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cancer Care Manitoba, Winnepeg, Manitoba
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
- Czechia (3):
  - Nemocnice odd. Onkologie, České Budějovice
  - Pneumologicka klinika 1. LF UK, Praha-6-Veleslavin
  - Klinika pneumologie a hrudni chirurgie 3.LF, Praha-8
- France (4):
  - Centre Hospitalier General de Belfort, Belfort, Cedex
  - Centre Hospitalier Francois Maillot, Briey, Cedex
  - Institut Jean Godinot, Reims, Cedex
  - Centre Hospitalier Intercommunal de la Haute-Saone, Vesoul, Cedex
- Greece (7):
  - University Hospital of Alexandroupolis, Dragana, Alexandroupolis
  - University General Hospital of Heraklion, Heraklion, Crete
  - 1st Pulmonary Clinic of G. Papanikolaou Hospital, Exochi, Thessaloniki
  - 2nd Pulmonary Clinic of G. Papanikolaou Hospital, Exochi, Thessaloniki
  - 6th Pneumonology Department, Sotiria Hospital for Diseases of the Chest, Athens
  - 7th Pneumonology Clinic, Sotiria Hospital for Diseases of the Chest, Athens
  - University Hospital of Patras, Rio
- Hungary (4):
  - Semmelweis University Department of Pulmonology, Budapest
  - Fovarosi Onkormanyzat Uzsoki utcai, Korhaza, Budapest
  - Koranyi National Institute for Pulmonology, Budapest
  - Csongrad Megyei Onkormanyzat Mellkasi, Deszk
- Israel (7):
  - Barzilai Medical Centre, Ashkelon
  - Hadassah Medical Center, Jerusalem
  - Meir Hospital, Kfar Saba
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sovrasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Ẕerifin
- Poland (5):
  - Regionalne Centrum Onkologii, Bialystok
  - Akademii Medycznej w Gdansku, Gdansk
  - Centrum Onkologii Instytut im. M. Sklodowskiej-Curie, Krakow
  - Wielkopolskie Centrum Chorob Pluc I Gruzlicy, Poznan
  - Instytut Gruzlicy i Chorob Pluc, Warsaw
- Russia (9):
  - Arkhangelsk Regional Oncology Center, Arkhangelsk
  - City Oncology Clinical Center, Moscow
  - Russian Oncology Research Center n.a. Blokhin, Moscow
  - Research Institute of Oncology n.a. Hertzen, Moscow
  - Central Clinical Hospital n.a. Semashko, Moscow
  - City Oncology Hospital #62, Moscow
  - City Oncology Center, Saint Petersburg
  - St. Petersburg Pavlov State Medical University, Saint Petersburg
  - Research Institute of Oncology n.a. Petrov, Saint Petersburg
- United Kingdom (6):
  - Aberdeen Royal Infirmary, Foresterhill, Aberdeen
  - Bristol Hematology and Oncology Centre, Bristol, England
  - Leicester Royal Infirmary, Leicester, England
  - Guys & St. Thomas' Cancer Centre, London, England
  - Chelsea & Westminster Hospital, London, England
  - University of Edinburgh, Edinburgh, Scotland

REFERENCES:
- See also: Related Info — http://www.Ligand.com